CLINICAL TRIAL: NCT02087709
Title: Effect of Hypocaloric Diet on Biomarkers of Metabolic Profile, Insulin Resistance and Body Composition in Women With Metabolic Syndrome
Brief Title: Effect of Low-calorie Diet on Serum Lipids, Adipokines, Insulin Resistance and Also Body Composition in Women With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Rio de Janeiro State University (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Grazielle Vilas Boas Huguenin, Mrs, Universidade Federal do Rio de Janeiro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0535.0.000.325-08; U1111-1154-4418 (Other: Universal trial number)
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Weight Loss; Insulin Resistance; Adipokines
MeSH Terms: conditions — Weight Loss; Insulin Resistance | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low-calorie diet (Experimental): The subjects were prescribed a daily energy intake 500 kcal lower than the estimated energy requirement.
  Interventions: Other: Low-calorie diet

INTERVENTIONS:
Other: Low-calorie diet

SUMMARY:
The purpose of this study is to evaluate the effect of a hypocaloric diet on biomarkers associated with insulin resistance, metabolic profile and body composition in women with Metabolic Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 30-34.9 kg/m2, diagnostic of metabolic syndrome based on National Cholesterol Education Panel ATPIII (2002)

Exclusion Criteria:

* Diabetes mellitus, non-treated thyroid disease, treatment with lipid-lowering drugs and glucocorticoids or weight loss treatment within the previous 3 months.

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Weight | Change from baseline at 3rd month
  Change from baseline weight (Kg) at 3rd month.

SECONDARY OUTCOMES:
Insulin resistance markers | Change from baseline at 3rd month
  Change from baseline fasting glucose and insulin, homeostasis model assessment-insulin resistance and quantitative insulin sensitivity check index at 3rd month, samples were stored at -20 degrees.

OTHER OUTCOMES:
Adipokines | Change from baseline at 3rd month
  The change from baseline leptin and adiponectin at 3rd month, samples were stored at -20 degrees

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil